CLINICAL TRIAL: NCT04703114
Title: Study of the Immunological and Virological Response of Patients Infected With SARS-CoV-2 and Presenting an Asymptomatic or Pauci-symptomatic Form
Brief Title: Study of the Immunological and Virological Response of Patients With COVID-19 and Presenting an Asymptomatic or Pauci-symptomatic Form (AMBUCOV)
Acronym: AMBUCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fonds IMMUNOV (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMBUCOV; 2020-A03102-37 (Other: ID-RCB)
Record Dates: First submitted 2020-11-30; First posted 2021-01-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19; SARS-CoV-2
Keywords: Covid19; SARS-CoV-2; Immunology
MeSH Terms: conditions — COVID-19 | interventions — Blood Cell Count; Blood Specimen Collection; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symptomatic (Experimental): 40 symptomatic patients to COVID-19 infection
  Interventions: Diagnostic Test: Blood count; Diagnostic Test: Blood collection; Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Saliva samples; Diagnostic Test: Faeces samples; Genetic: Genetic blood collection; Other: Data collection
- Asymptomatic (Experimental): 40 asymptomatic patients to COVID-19 infection
  Interventions: Diagnostic Test: Blood count; Diagnostic Test: Blood collection; Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Saliva samples; Diagnostic Test: Faeces samples; Genetic: Genetic blood collection; Other: Data collection

INTERVENTIONS:
Diagnostic Test: Blood count — Blood count at each visit
Diagnostic Test: Blood collection — Blood collection to understanding of the immunological profile at each visit
Diagnostic Test: Nasopharyngeal swab — Research of SARS-CoV-2 infection in nasopharyngeal swab by RT-PCR at day 8 and day 15
Diagnostic Test: Saliva samples — Research of SARS-CoV-2 infection in saliva samples at each visit (excepted inclusion)
Diagnostic Test: Faeces samples — Research of SARS-CoV-2 infection in faeces samples at day 3, day 15 and day 90
Genetic: Genetic blood collection — Collection to further research at each visit
Other: Data collection — Demographics, symptoms, biological constants

SUMMARY:
The purpose of this study is to describe the immunological and virological response of patients infected with CoV-2-SARS and presenting an asymptomatic or mildly symptomatic form, in particular the innate and adaptive response as well as the virological clearance kinetics.

The research hypothesis is that patients with an ambulatory form of SARS-CoV-2 infection, whether asymptomatic or mildly symptomatic, are able to mount an innate and adaptive immunological response capable of rapidly clearing the virus, in contrast to severe forms in which an early deficit of type 1 IFN response has been demonstrated, possibly responsible for a defect in the control of viral replication in the blood.

DETAILED DESCRIPTION:
A new coronavirus (SARS-CoV-2) was identified in December 2019 in the Wuhan region of China and is currently causing a global pandemic.

The disease, named COVID-19, causes an influenza syndrome associated with respiratory signs, but there are also asymptomatic and pauci-symptomatic forms. Approximately 2 to 3% of patients, primarily patients with pre-existing chronic diseases and the elderly, develop a very severe form responsible for an acute respiratory distress syndrome (ARDS) that can lead to death.

It has been shown that patients with a severe and critical form had an impaired type 1 interferon response, with decreased plasma levels of IFN-alpha2 in the most severe patients compared to hospitalized patients with a moderate form, and undetectable levels of IFN-beta. This lack of type 1 IFN response was associated with greater viral persistence in the blood and an exaggerated inflammatory response mediated primarily by the NF-kB pathway.

Almost all studies published to date on immune system disruption during CoV-2-SARS infection included mainly hospitalized patients requiring oxygen therapy due to their severity, assessed at the time of clinical worsening.

Thus, there is no or little data on immunological response profiles, particularly on type 1 IFN response but also on other aspects of the immunological response (adaptive cellular and humoral immunity), and its relationship with viral clearance kinetics during ambulatory forms of SARS-CoV-2 infection, whereas these forms represent more than 95% of the clinical forms.

The asymptomatic and pauci-symptomatic forms managed on an outpatient basis represent the most common form of CoV-2-SARS infection, with a favourable outcome in almost all cases.

A better description and understanding of the immunological profile, including type 1 IFN response and viral clearance kinetics in saliva, blood and feces, during asymptomatic and mild clinical forms will allow the identification of the major players in the immune response against SARS-CoV-2, and thus better define the responses that are lacking in severe patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Nasopharyngeal PCR positive for SARS-CoV-2 within 48 hours prior to inclusion in the study protocol, carried out in one of the participating outpatient screening centers
* Symptomatic patients (nasopharyngeal screening positive due to suggestive symptoms) or asymptomatic (nasopharyngeal screening positive due to screening after contact with a positive subject)
* Patients who have been informed and signed the consent
* Pregnant and breastfeeding women who may be included in the study.

Exclusion Criteria:

* Patients with criteria for hospitalization at the time of diagnosis (seriousness criteria, impossibility of staying at home)
* Non-consent or inability to obtain consent,
* Patient with dementia or not authorized, for psychiatric reasons or intellectual failure, to receive information on the protocol and to give informed consent,
* Patient under guardianship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Interferon response | Up to 90 days
  Concentration of type I, type II and type III Interferon in peripheral blood

SECONDARY OUTCOMES:
Immunology : cytokines | Up to 90 days
  Concentration of IL-6, TNF-alpha, IL-8, calprotectin in peripheral blood
Immunology : cell population | Up to 90 days
  Proportions of monocytes, B cells and T cells in peripheral blood
Immunology : proteins | Up to 90 days
  Concentration of anaphylatoxins C3a and C5a in peripheral blood
Immunology : pathways | Up to 90 days
  Screening for genetic mutations involved in the interferon pathway
Immunology : antibody response | Up to 90 days
  Concentration of antibodies directed against spike protein and nucleocapsids
Virology : Nasopharyngeal Viral clearance kinetics | Up to 90 days
  Viral clearance kinetics in nasopharyngeal samples
Virology : Saliva Viral clearance kinetics | Up to 90 days
  Viral clearance kinetics in saliva
Virology : faeces viral clearance kinetics | Up to 90 days
  Viral clearance kinetics in faeces
Virology : peripheral blood viral clearance kinetics | Up to 90 days
  Viral clearance kinetics in peripheral blood
Virology : sequencing | Up to 90 days
  Analysis of virus mutations, especially of the gene encoding spike protein

CONTACTS AND LOCATIONS:
Overall Officials: Solen KERNEIS, Doctor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lingas G, Planas D, Pere H, Porrot F, Guivel-Benhassine F, Staropoli I, Duffy D, Chapuis N, Gobeaux C, Veyer D, Delaugerre C, Le Goff J, Getten P, Hadjadj J, Bellino A, Parfait B, Treluyer JM, Schwartz O, Guedj J, Kerneis S, Terrier B. Neutralizing Antibody Levels as a Correlate of Protection Against SARS-CoV-2 Infection: A Modeling Analysis. Clin Pharmacol Ther. 2024 Jan;115(1):86-94. doi: 10.1002/cpt.3069. Epub 2023 Oct 20. PMID 37795693
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Hadjadj J, Yatim N, Barnabei L, Corneau A, Boussier J, Smith N, Pere H, Charbit B, Bondet V, Chenevier-Gobeaux C, Breillat P, Carlier N, Gauzit R, Morbieu C, Pene F, Marin N, Roche N, Szwebel TA, Merkling SH, Treluyer JM, Veyer D, Mouthon L, Blanc C, Tharaux PL, Rozenberg F, Fischer A, Duffy D, Rieux-Laucat F, Kerneis S, Terrier B. Impaired type I interferon activity and inflammatory responses in severe COVID-19 patients. Science. 2020 Aug 7;369(6504):718-724. doi: 10.1126/science.abc6027. Epub 2020 Jul 13. PMID 32661059
- [Background] Lucas C, Wong P, Klein J, Castro TBR, Silva J, Sundaram M, Ellingson MK, Mao T, Oh JE, Israelow B, Takahashi T, Tokuyama M, Lu P, Venkataraman A, Park A, Mohanty S, Wang H, Wyllie AL, Vogels CBF, Earnest R, Lapidus S, Ott IM, Moore AJ, Muenker MC, Fournier JB, Campbell M, Odio CD, Casanovas-Massana A; Yale IMPACT Team; Herbst R, Shaw AC, Medzhitov R, Schulz WL, Grubaugh ND, Dela Cruz C, Farhadian S, Ko AI, Omer SB, Iwasaki A. Longitudinal analyses reveal immunological misfiring in severe COVID-19. Nature. 2020 Aug;584(7821):463-469. doi: 10.1038/s41586-020-2588-y. Epub 2020 Jul 27. PMID 32717743